CLINICAL TRIAL: NCT02180750
Title: An Evaluation of a Psychosocial Intervention for Orphans With HIV Infection: a Phase II Randomised Controlled Trial of Memory Work Therapy at PASADA, Tanzania
Brief Title: Phase II Randomised Controlled Trial of Memory Work Therapy at PASADA, Tanzania
Acronym: MWT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pastoral Activities and Service for AIDS Dar-Es-Salaam Archdiocese (Other)
Collaborators: University of Cape Town (Other); King's College London (Other)
Responsible Party: Principal Investigator, Elvis Joseph Miti, Social Worker, Pastoral Activities and Service for AIDS Dar-Es-Salaam Archdiocese
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MWT01
Record Dates: First submitted 2014-06-24; First posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: HIV
Keywords: Children; HIV; orphans
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: Memory Work Therapy (Experimental): Residential week intervention consisting of memory box, memory book, tree of life, Active Citizen book, all activities facilitated.
  Interventions: Other: Memory Work Therapy
- Control: standard care (Active Comparator): Usual care services.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Memory Work Therapy
  Arms: Intervention: Memory Work Therapy
Other: Standard care — Pediatric clinic, ART
  Arms: Control: standard care

SUMMARY:
Memory Work Therapy (MWT) has been developed to improve psycho-social outcomes for children living with HIV who are orphaned. This phase 2 trial aims to determine whether attending the intervention improves outcomes compared to standard care. We aim to test the hypothesis that attendance at MWT improves psychological symptoms, self-esteem, emotional and behavioural difficulties, and self-efficacy compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14-18 years
* HIV positive
* Orphaned
* Naïve to the intervention

Exclusion Criteria:

* Adults
* Children under 14
* HIV negative
* Parent(s) living
* Previously attended the intervention

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-07 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Change: Brief Symptom Inventory | T0( study entry), T1 (2 weeks), T2 (6 weeks)
  The BSI measures psychological symptom patterns

SECONDARY OUTCOMES:
Change: Rosenberg Self-Esteem Scale | T0 (study entry), T1 (2 weeks), T2 (6 weeks)
  A measure of self esteem
Change: Goodman's strengths and difficulties questionnaire | T0 (study entry), T1 (2 weeks) T2 (6 weeks)
  Measures mental health in children and young people
Change: Self-efficacy questionnaire for children | T0 (study entry), T1 (2 weeks), T2 (6 weeks)
  measure emotional and social self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- PASADA, Temeke, Tanzania

REFERENCES:
- [Derived] Harding R, Wei G, Gwyther L, Miti E. Improving psychological outcomes for orphans living with HIV in Tanzania through a novel intervention to improve resilience: findings from a pilot RCT. AIDS Care. 2019 Mar;31(3):340-348. doi: 10.1080/09540121.2018.1533630. Epub 2018 Oct 17. PMID 30332895